CLINICAL TRIAL: NCT03074136
Title: Application Success of Photodynamic Therapy and Diode Laser During Endodontic Therapy of Young Permanent Teeth
Brief Title: Application of Photodynamic Therapy and Diode Laser for Endodontic Therapy of Young Permanent Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association of Paediatric and Preventive Dentists of Serbia (Other)
Responsible Party: Principal Investigator, Dejan Markovic, Professor, Association of Paediatric and Preventive Dentists of Serbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36/8
Record Dates: First submitted 2017-02-11; First posted 2017-03-08 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Teeth, Endodontically-Treated
Keywords: photodynamic therapy; diode laser; immature permanent teeth; endodontic therapy
MeSH Terms: conditions — Tooth, Nonvital | interventions — Lasers, Semiconductor; Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photodinamic therapy (Experimental): Chemomechanical preparation will be completed by hand instruments, with minimal instrumentation, and usage of sodium hypochlorite with minimal bactericidal concentration (0.5%, pH 12), on room temperature (21 degree Celsius). After that, HELBO treatment (Helbo Photodynamic System, Bredent, Senden, Germany) will be applied.
  Interventions: Device: Photodinamic therapy; Drug: 0.5% Sodium hypochlorite
- Diode laser (Experimental): Chemomechanical preparation will be completed by hand instruments, with minimal instrumentation, and usage of sodium hypochlorite with minimal bactericidal concentration (0.5%, pH 12), on room temperature (21 degree Celsius). After that high power diode laser therapy will be applied by using Epic diode laser (Biolase® Technology, Inc., San Clemente, CA, USA).
  Interventions: Device: Diode laser; Drug: 0.5% Sodium hypochlorite
- 0.5% Sodium hypochlorite (Experimental): Chemomechanical preparation will be completed by hand instruments, with minimal instrumentation, and usage of sodium hypochlorite with minimal bactericidal concentration (0.5%, pH 12), on room temperature (21 degree Celsius).
  Interventions: Drug: 0.5% Sodium hypochlorite

INTERVENTIONS:
Device: Photodinamic therapy — Dentin sealant (HELBO® Endo Seal, Bredent, Senden, Germany) will be applied over the crown area and light cured. The root canals will be filled with the phenothiazine chloride (HELBO® Endo Blue, Bredent, Senden, Germany), agitated with a size 15K-file and left in the canal for 2 min. After this time, the root canals will be rinsed with distilled water to remove the excess of the photosensitizer, dried with paper points. The disposable 450 µm fiberoptic tip (3D HELBO® Endo Probe, Bredent, Senden, Germany) will be placed in the apical portion of the root canal at the point where resistance to the fiber will be felt, and root canal will be irradiated with HELBO® TheraLite Laser (λ = 660 nm, power = 100 mW) for 60 s (total energy, 6 J) in a continuous wave mode.
  Other Names: PDT
  Arms: Photodinamic therapy
Device: Diode laser — High-power diode laser therapy will be applied by using Epic diode laser (Biolase® Technology, Inc., San Clemente, CA, USA) with settings determined in laboratory researches (λ = 940 nm, maximal power 10W).
  Other Names: High-power diode laser
  Arms: Diode laser
Drug: 0.5% Sodium hypochlorite — Chemomechanical preparation will be completed by hand instruments, with minimal instrumentation, and usage of sodium hypochlorite with minimal bactericidal concentration (0.5%, pH 12), on room temperature (21 degrees Celsius).
  Other Names: 0.5% NaOCl

SUMMARY:
The pulp necrosis of permanent immature teeth implies the interruption of the root formation and apical closure. Diode lasers have been used in many areas of dentistry, with tendency of good results in canal and dentine disinfection. The bactericidal effect of high-power lasers is based on dose dependent heat generation. Its antimicrobial effectiveness against diverse microorganisms has already been demonstrated. Photodynamic therapy (PDT) is a two-step therapeutic approach starting with the application of a photosensitizing agent and followed by irradiation with light energy that is spectrally matched to activate the drug. The balance between disinfection and the creation of an intracanal microenvironment conducive for the proliferation of stem cells requires further investigation. Aims of study are to compare the time required to obtain the clinical healing and the disappearance of clinical symptoms, and absence of periapical radiolucency, by using PDT and diode laser, with standard disinfection alone; to assess specificity of microbial load in permanent immature teeth, and root canal disinfection ability of PDT and diode laser, in compare with standard disinfection alone.

DETAILED DESCRIPTION:
Background and Significance The pulp necrosis of permanent immature teeth implies the interruption of the root formation and apical closure. It is then necessary to implement a therapy to induce a calcified barrier at the apical end of the root. The endodontic management of permanent immature teeth is fraught with challenges. Although treatment modalities for vital pulp therapy in these teeth provide long-term favorable outcome, the outcomes from the treatment of pulp necrosis and apical periodontitis are significantly less predictable. Key role of microorganisms in the causing and development of pulpal and periapical diseases have been demonstrated, and their presence in the canal at the time of definitive filling has negative effect on success of the therapy. However, the specificity of microbial load of immature permanent teeth is not completely investigated, nor the influence of the disinfection protocols on treatment success.

Available procedures rely heavily on root canal chemical disinfection of the root canal system, with minimal mechanical instrumentation. Sodium hypochlorite (NaOCl) in different concentrations is the most accepted solution for disinfection of root canal in endodontic. Despite common usage, impossibility of NaOCl to completely disinfect root canal has been noticed. Traditionally, irrigants and medicaments have been chosen for their maximum antimicrobial effect without consideration for their effects on stem cells and the dentinal microenvironment. The balance between disinfection and the creation of an intracanal microenvironment conducive for the proliferation of stem cells requires further investigation. This requires the interpretation of preclinical studies, and this level of evidence should be increased by randomized controlled clinical studies.

Diode lasers have been used in many areas of dentistry, with tendency of good results in canal and dentine disinfection. The bactericidal effect of high-power lasers is based on dose dependent heat generation. Its antimicrobial effectiveness against diverse microorganisms has already been demonstrated.

Photodynamic therapy (PDT) is a two-step therapeutic approach starting with the application of a photosensitizing agent and followed by irradiation with light energy that is spectrally matched to activate the drug. Because its high antibacterial potential, usage of photodynamic therapy as advance to standard protocol in root canal disinfection have been suggested. Studies showed positive effect of photodynamic therapy in the reduction of microbial load in root canal treatment. When a photoactive compound is applied in the root canal system, it is taken up by residual bacteria in the main canals, isthmuses, lateral canals and dentinal tubules. It is also possible that this compound may escape into the periapical tissues. During PDT, light will excite the drug in bacteria within the root canal, but could also potentially affect the apical stem cells that have taken up the drug. Therefore, it is important to determine the therapeutic window whereby host cells are left intact.

Several studies showed wide-ranging spectra of desirable effects of low level power laser (LLLT) on biological tissue. It has been reported to increase cell functional activity, induce cell proliferation, lowers inflammation, releasing of endorphins, thus having analgetic effect. Furthermore, it has been shown that irradiation with a LLLT following photosensitization with phenothiazine chloride had no negative effect on the growth and differentiation of human osteoblastic cells, and did not counteract the biostimulatory effect induced by LLLT. There were no statistically significant differences in the growth and differentiation behavior between the two study groups. Further investigations of PDT on dental stem cells are needed to determine possible biostimulative effect on proliferation and differentiation, and thereby contribute to root development of non-vital permanent immature teeth. Prolonged treatment of young permanent teeth increases possibility of treatment failure. Involvement of a method that could help healing process is desirable.

ELIGIBILITY:
Inclusion criteria

* a non-vital permanent immature single rooted tooth
* primary endodontic infection
* 6 - 18 years old
* written informed consent obtained from each parent and child

Exclusion criteria

* uncontrolled diabetes mellitus,
* immunosuppression,
* severe asthma
* usage of antibiotics, anti-inflammatory, corticosteroid, or immunosuppressive therapy during the last 6 months
* need for antibiotics at current endodontic therapy
* need for antibiotics in prophylaxis of systematic disease before endodontic therapy
* periodontal diseases
* impossible adequate isolation of the tooth

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Number of teeth without viable bacteria load in root canal after Photodynamic therapy and Diode laser in endodontic therapy | 6 months
  Number of teeth without viable bacteria load after treatment in all experimental groups, will be determined. Microbiological samples from the root canals will be collected immediately after the accessing the canal, following endodontic treatment, and after the laser procedure in adequate groups (Photodynamic therapy or Diode laser). Samples from the root canals will be cultivated in conditions suitable for growth of anaerobes and facultative anaerobes.

SECONDARY OUTCOMES:
Number of teeth with periapical healing 6 months after treatment, assessed by periapical index (PAI) | 6 months
  Number of teeth with periapical healing 6 months after treatment, will be determined by PAI score index, in all experimental groups. Teeth will be categorized in five groups depending of PAI score: (1) normal periapical structure; (2) small changes in bone structure; (3) changes in bone structure with some mineral loss; (4) periodontitis with well-defined radiolucent area; and (5) severe periodontitis with exacerbating features.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diogenes AR, Ruparel NB, Teixeira FB, Hargreaves KM. Translational science in disinfection for regenerative endodontics. J Endod. 2014 Apr;40(4 Suppl):S52-7. doi: 10.1016/j.joen.2014.01.015. PMID 24698694
- [Background] Siqueira JF Jr, Rocas IN. Clinical implications and microbiology of bacterial persistence after treatment procedures. J Endod. 2008 Nov;34(11):1291-1301.e3. doi: 10.1016/j.joen.2008.07.028. Epub 2008 Sep 17. PMID 18928835
- [Background] Shabahang S, Pouresmail M, Torabinejad M. In vitro antimicrobial efficacy of MTAD and sodium hypochlorite. J Endod. 2003 Jul;29(7):450-2. doi: 10.1097/00004770-200307000-00006. PMID 12877261
- [Background] Waltimo T, Trope M, Haapasalo M, Orstavik D. Clinical efficacy of treatment procedures in endodontic infection control and one year follow-up of periapical healing. J Endod. 2005 Dec;31(12):863-6. doi: 10.1097/01.don.0000164856.27920.85. PMID 16306819
- [Background] Pearson GJ, Schuckert KH. The role of lasers in dentistry: present and future. Dent Update. 2003 Mar;30(2):70-4, 76. doi: 10.12968/denu.2003.30.2.70. PMID 12705027
- [Background] Gutknecht N, Franzen R, Schippers M, Lampert F. Bactericidal effect of a 980-nm diode laser in the root canal wall dentin of bovine teeth. J Clin Laser Med Surg. 2004 Feb;22(1):9-13. doi: 10.1089/104454704773660912. PMID 15117481
- [Background] Soukos NS, Chen PS, Morris JT, Ruggiero K, Abernethy AD, Som S, Foschi F, Doucette S, Bammann LL, Fontana CR, Doukas AG, Stashenko PP. Photodynamic therapy for endodontic disinfection. J Endod. 2006 Oct;32(10):979-84. doi: 10.1016/j.joen.2006.04.007. Epub 2006 Jul 13. PMID 16982278
- [Background] Chrepa V, Kotsakis GA, Pagonis TC, Hargreaves KM. The effect of photodynamic therapy in root canal disinfection: a systematic review. J Endod. 2014 Jul;40(7):891-8. doi: 10.1016/j.joen.2014.03.005. Epub 2014 May 2. PMID 24935531
- [Background] Xu Y, Young MJ, Battaglino RA, Morse LR, Fontana CR, Pagonis TC, Kent R, Soukos NS. Endodontic antimicrobial photodynamic therapy: safety assessment in mammalian cell cultures. J Endod. 2009 Nov;35(11):1567-72. doi: 10.1016/j.joen.2009.08.002. Epub 2009 Sep 20. PMID 19840649
- [Background] Toomarian L, Fekrazad R, Tadayon N, Ramezani J, Tuner J. Stimulatory effect of low-level laser therapy on root development of rat molars: a preliminary study. Lasers Med Sci. 2012 May;27(3):537-42. doi: 10.1007/s10103-011-0935-9. Epub 2011 May 26. PMID 21614480
- [Background] Martens LC. Laser physics and a review of laser applications in dentistry for children. Eur Arch Paediatr Dent. 2011 Apr;12(2):61-7. doi: 10.1007/BF03262781. PMID 21473835
- [Background] Stein E, Koehn J, Sutter W, Schmidl C, Lezaic V, Wendtlandt G, Watzinger F, Turhani D. Phenothiazine chloride and soft laser light have a biostimulatory effect on human osteoblastic cells. Photomed Laser Surg. 2009 Feb;27(1):71-7. doi: 10.1089/pho.2008.2265. PMID 19196108
- [Background] Juric IB, Plecko V, Panduric DG, Anic I. The antimicrobial effectiveness of photodynamic therapy used as an addition to the conventional endodontic re-treatment: a clinical study. Photodiagnosis Photodyn Ther. 2014 Dec;11(4):549-55. doi: 10.1016/j.pdpdt.2014.10.004. Epub 2014 Oct 24. PMID 25461966